CLINICAL TRIAL: NCT01984294
Title: A Phase 2, Randomized, Open-Label Study of Sofosbuvir/Ledipasvir Fixed-Dose Combination With Ribavirin or GS-9669 250 mg or GS-9669 500 mg in Naive or Treatment-Experienced Cirrhotic Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination With Ribavirin or GS-9669 in Subjects With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0133
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2015-04

CONDITIONS: Chronic HCV Infection
Keywords: HCV genotype 1; HCV; Sustained Virologic Response; Direct-Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Open Label; Sofosbuvir; Treatment-Naive; Protease Inhibitors; PI; Treatment experienced; Cirrhotic
MeSH Terms: interventions — Ribavirin; GS-9669

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LDV/SOF+RBV (Experimental): Participants will receive LDV/SOF plus RBV for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF + GS-9669 250 mg (Experimental): Participants will receive LDV/SOF plus GS-9669 250 mg for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: GS-9669
- LDV/SOF + GS-9669 500 mg (Experimental): Participants will receive LDV/SOF plus GS-9669 500 mg (2 x 250 mg) for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: GS-9669

INTERVENTIONS:
Drug: LDV/SOF — Ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5885
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
  Arms: LDV/SOF+RBV
Drug: GS-9669 — GS-9669 tablet(s) administered orally once daily
  Arms: LDV/SOF + GS-9669 250 mg; LDV/SOF + GS-9669 500 mg

SUMMARY:
This study will evaluate the antiviral efficacy of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) plus ribavirin (RBV) or LDV/SOF plus GS-9669 in treatment-naive or treatment-experienced participants with chronic genotype 1 hepatitis C virus (HCV) infection. A total of 90 participants are planned to be enrolled in the study for 8 weeks of treatment, approximately 60 having had prior treatment with a regimen containing pegylated interferon (PEG) and RBV for ≥ 12 weeks. Randomization will be stratified by treatment-naive versus treatment-experienced and by HCV genotype (1a versus 1b).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, with chronic genotype 1 HCV infection
* Documented HCV treatment-naïve or treatment-experienced subjects who failed previous PEG+RBV regimen
* HCV RNA > 10,000 IU/mL at Screening
* Presence of compensated cirrhosis
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hyland, DPhil, Study Director — Gilead Sciences
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 1 study site in the United States. The first participant was screened on 29 October 2013. The last study visit occurred on 18 July 2014.
Pre-assignment Details: 117 participants were screened.
Groups:
- LDV/SOF+RBV: Ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg fixed-dose combination (FDC) tablet once daily plus ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) in a divided daily dose for 8 weeks
- LDV/SOF+GS-9669 250 mg: LDV/SOF 90/400 mg FDC tablet plus GS-9669 (1 x 250 mg) tablet once daily for 8 weeks
- LDV/SOF+GS-9669 500 mg: LDV/SOF 90/400 mg FDC tablet plus GS-9669 (2 x 250 mg) tablets once daily for 8 weeks
Period: Overall Study
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Started | 35 | 32 | 34
Completed | 31 | 29 | 27
Not Completed | 4 | 3 | 7
Not completed — Randomized but Never Treated | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 2 | 6
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug.
Groups:
- LDV/SOF+RBV: LDV/SOF 90/400 mg FDC tablet once daily plus RBV tablets (1000 or 1200 mg daily based on weight) in a divided daily dose for 8 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg | Total
Number analyzed (Participants) | 35 | 32 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.8) | 57 (7.4) | 57 (9.3) | 57 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 12 | 35
  Male | 20 | 24 | 21 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2 | 0 | 4 | 6
  White | 32 | 32 | 28 | 92
  American Indian/ Alaska Native | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 13 | 12 | 39
  Not Hispanic or Latino | 21 | 19 | 21 | 61
HCV Genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes.
  participants
    Genotype 1a | 21 | 20 | 21 | 62
    Genotype 1b | 14 | 12 | 12 | 38
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 5 | 6 | 7 | 18
    CT | 16 | 23 | 19 | 58
    TT | 14 | 3 | 7 | 24
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (0.50) | 6.1 (0.63) | 6.0 (0.57) | 6.0 (0.56)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 14 | 9 | 12 | 35
  ≥ 800,000 IU/mL | 21 | 23 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Number analyzed (Participants) | 35 | 32 | 33
percentage of participants | 88.6 | 90.6 | 81.8

2. Primary Outcome: Percentage of Participants Permanently Discontinuing Any Study Drug Due to an Adverse Event
Time Frame: Up to 8 weeks
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Number analyzed (Participants) | 35 | 32 | 33
percentage of participants | 0 | 3.1 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 2, 4, 8, and 24 Weeks After Discontinuation of Therapy (SVR2, SVR4, SVR8, and SVR24)
Description: SVR2, SVR4, SVR8, and SVR24 was defined as HCV RNA < LLOQ at 2, 4, 8, and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 2, 4, 8, and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Number analyzed (Participants) | 35 | 32 | 33
percentage of participants
  SVR2 | 100.0 | 100.0 | 97.0
  SVR4 | 91.4 | 90.6 | 84.8
  SVR8 | 88.6 | 90.6 | 81.8
  SVR24 | 88.6 | 90.6 | 81.8

4. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 8 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Number analyzed (Participants) | 35 | 32 | 33
percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Number analyzed (Participants) | 35 | 32 | 33
percentage of participants | 11.4 | 9.4 | 18.2

ADVERSE EVENTS:
Time Frame: Up to 8 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- LDV/SOF+RBV: LDV/SOF 90/400 mg FDC tablet once daily plus RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks
Arm/Group | LDV/SOF+RBV | LDV/SOF+GS-9669 250 mg | LDV/SOF+GS-9669 500 mg
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/32 | 0/33
Other Adverse Events (participants affected / at risk) | 24/35 | 13/32 | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV (N=35) | LDV/SOF+GS-9669 250 mg (N=32) | LDV/SOF+GS-9669 500 mg (N=33)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV (N=35) | LDV/SOF+GS-9669 250 mg (N=32) | LDV/SOF+GS-9669 500 mg (N=33)
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 2 | 2 | 1
Influenza like illness (General disorders) | 2 | 1 | 1
Asthenia (General disorders) | 2 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 7
Dizziness (Nervous system disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years